CLINICAL TRIAL: NCT03070457
Title: Safety of an Early Discharge Protocol After Sleeve Gastrectomy. Randomised Clinical Trial
Brief Title: Safety of an Early Discharge Protocol After Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Amador Garci-a Ruiz de Gordejuela, MD, PhD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC007/17
Record Dates: First submitted 2017-02-24; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Morbid Obesity; Sleeve Gastrectomy; Early Discharge; Safety Issues
Keywords: bariatric surgery; sleeve gastrectomy; eras
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early discharge group (Experimental): Patients with a shorter hospital stay, 23 hours after surgery
  Interventions: Other: Early discharge
- Conventional discharge (Active Comparator): Patients with conventional protocol and 48-72 hours of hospital stay
  Interventions: Other: Conventional protocol

INTERVENTIONS:
Other: Early discharge — Patients randomised to early discharge or not
  Arms: Early discharge group
Other: Conventional protocol — Discharge as usually done 48-72 hours after surgery
  Arms: Conventional discharge

SUMMARY:
Evaluate the safety and efficacy of an early discharge protocol (23 hours, overnight stay) after scheduled sleeve gastrectomy.

DETAILED DESCRIPTION:
This study aims to demonstrate that a shorter hospital stay after sleeve gastrectomy is as safe and useful as conventional protocol with 48-36 hours of stay. We consider that an adequate patient information and support will facilitate this shorter stay

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for Sleeve gastrectomy
* BMI 35 to 50
* ASA I to III
* Conventional address close to our Hospital
* Laparoscopic surgery
* Accompanying person after discharge
* Availability for a smart phone

Exclusion Criteria:

* ASA IV
* Revisional Surgery
* Conversion to laparotomy
* ICU Admission after surgery
* Insulin dependent Diabetes Mellitus
* Surgery finishing after 3 pm

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Readmissions rate | 1 month
  No hospital admissions after surgery

SECONDARY OUTCOMES:
Morbidity rate | 1 month
  Number of postoperative complications
Chronogram for complications after surgery | 1 month
  Detailed timing of appearance
Quality of life | 1 month
  BAROS questionnaire
Patients agreement to the protocol | 1 month
  Specific survey created ad hoc

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided